CLINICAL TRIAL: NCT05817734
Title: Longitudinal Collection of Observational Clinical and Lifestyle Data
Brief Title: Human Phenotype Project Study Protocol
Status: Recruiting | Type: Observational
Sponsor: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Eran Segal, Prof. Eran Segal, PI at the department of computer science and applied math, Weizmann Institute of Science
Other Study IDs: 1789-1
Record Dates: First submitted 2023-01-31; First posted 2023-04-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Adult Disease
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and stool sampls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective study aimed at recruiting 30,000 individuals, aged 40-70 years old, and following them longitudinally for 25 years with repeated measurements. The basic follow-up frame will include a visit to the Clinical Test Center (CTC) every two years and a phone interview every other year (on uneven years). Sample collection and biobanking will be performed every two years and online questionnaires will be filled out on an annual basis.

The primary goals are to study the variation observed across different individuals in disease susceptibility, clinical phenotypes, and therapeutic responses. The study aims at studying the complex interplay and relative contribution of different omics, physiological characteristics and lifestyle on disease pathogenesis and progression and to evaluate how these effects are mediated.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18+, males and females.

Exclusion Criteria:

* Pregnancy.
* Mentally disabled or in general legally non-competent.
* Prisoner or soldier. Soldiers: mandatory service only
* Active cancer
* Fertility Treatments (current)
* Hepatitis ( B, C), chronic or acute
* HIV
* Liver cirrhosis
* Dialysis
* Unstable medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General volunteering population who can freely register for the study.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2045-12-31 (Estimated); Study Completion 2045-12-31 (Estimated)

PRIMARY OUTCOMES:
Adult disease | 25 years
  Development of medical conditions based on participant's self-reporting coded to ICD11.

CONTACTS AND LOCATIONS:
Locations (1):
- Weizmann institute of science, Rehovot, Israel

REFERENCES:
- [Derived] Rein M, Elkan M, Godneva A, Dolev NC, Segal E. Sex-specific dietary habits and their association with weight change in healthy adults. BMC Med. 2024 Nov 6;22(1):512. doi: 10.1186/s12916-024-03730-3. PMID 39501340